CLINICAL TRIAL: NCT06283394
Title: AHA (American Heart Association) Health Care x Food Penn Medicine Food Market Study
Brief Title: Penn Medicine Food Market Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 854803
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Usual Care (No Intervention): Participants in the usual care arm will not receive weekly subsidies on Instacart, and they will not receive any modifications to the virtual storefront on Instacart. They will have access to the standard Instacart platform and Instacart + memberships with a $5 per week to cover service and delivery fees and coverage of delivery tips for 3 months.
- Non Choice Architecture (Arm A) (Experimental): Arm A will receive a $160 subsidy per month for 3 months to be used on healthy foods (fruits and vegetables, whole grains, etc.). They will see the Instacart storefront without choice architecture manipulation and will see the discount applied at checkout. They will have Instacart + memberships for 3 months.
  Interventions: Behavioral: Fresh Funds
- Choice Architecture (Arm B) (Experimental): Arm B will receive a $160 subsidy per month for 3 months to be used on healthy foods (fruits and vegetables, whole grains, etc.). They will see a storefront with choice architecture manipulation (healthy items for diabetics appear first and less healthy items are less visible) and will see the discount applied at checkout. They will have Instacart + memberships for 3 months.
  Interventions: Behavioral: Storefront Choice Architecture; Behavioral: Fresh Funds
- Non Choice Architecture + Loss Framing (Arm C) (Experimental): Arm C will receive a $160 subsidy per month for 3 months to be used on produce.They will see the usual Instacart storefront and will see the discount applied at checkout. They will also receive text messages detailing how much of their $160 subsidy is left (beginning of weeks 1, 2, 3, and 4 and following the end of the month). They will have Instacart + memberships.
  Interventions: Behavioral: Fresh Funds; Behavioral: Loss Framing
- Choice Architecture + Loss Framing (Arm D) (Experimental): Arm D will receive a $160 subsidy per month for 3 months to be used on produce. They will see a storefront with choice architecture manipulation (healthy items for diabetics appear first and less healthy items are less visible) and will see the discount applied at checkout. They will also receive text messages detailing how much of their $160 subsidy is left (as in arm C). They will have Instacart + memberships.
  Interventions: Behavioral: Storefront Choice Architecture; Behavioral: Fresh Funds; Behavioral: Loss Framing

INTERVENTIONS:
Behavioral: Storefront Choice Architecture — An Instacart storefront with choice architecture manipulation (healthy items for diabetics appear first and less healthy items are less visible)
  Arms: Choice Architecture (Arm B); Choice Architecture + Loss Framing (Arm D)
Behavioral: Fresh Funds — The treatment groups will each receive a $160 subsidy per month for 3 months to be used on produce through Instacart.
  Arms: Choice Architecture (Arm B); Choice Architecture + Loss Framing (Arm D); Non Choice Architecture (Arm A); Non Choice Architecture + Loss Framing (Arm C)
Behavioral: Loss Framing — They will receive text messages detailing how much of their $160 subsidy is left (beginning of weeks 1, 2, 3, and 4 and following end of the month).
  Arms: Choice Architecture + Loss Framing (Arm D); Non Choice Architecture + Loss Framing (Arm C)

SUMMARY:
The goal of this interventional study is to test ways to improve the effectiveness of a healthy foods prescription program in increasing the purchase of healthy foods for patients who have both obesity (BMI >or= 30) and diabetes (last A1C>8 in the 90 days from data pull). The main questions it aims to answer are:

Aim 1: Examine feasibility and engagement among participants by assessing percent enrollment among those identified as eligible, rates of Instacart platform use, amount of the subsidy used each week, and amounts of healthy foods ordered.

Aim 2: Examine strategies to optimize the user experience of trial participation, including communication strategies and on-boarding, to increase uptake and engagement in this and subsequent studies.

Usual Care (Control): Participants in the usual care arm will not receive weekly subsidies on Instacart, and they will not receive any modifications to the virtual storefront on Instacart. They will have access to the standard Instacart platform and Instacart + memberships with $5 per week to cover service and delivery fees and delivery tips for 3 months.

Intervention Arms: The four treatment groups will also each receive a $160 subsidy per month for 3 months to be used on produce (fruits and vegetables).

DETAILED DESCRIPTION:
Patients who have both obesity (BMI >or= 30) and diabetes (last A1C>8 in the 90 days from time of data pull) will be recruited from specific Penn Medicine primary care practices. This patient list is curated based on the inclusion/exclusion criteria.

Participants in the control group will receive usual care (defined as access to the the virtual storefront without the choice architecture manipulation) but all study participants will receive a free Instacart+ membership for the 3 months they are a study participant and be given $20 per month to help cover the cost of additional delivery and service fees as well as tips for delivery drivers on Instacart. Participants in the intervention groups will in addition receive $160 per month in subsidies on Instacart. All arms will receive text messages and/or email messages from W2H 1x per week with a link to Instacart and different messaging depending on the study arm.

The main difference between the pilot intervention and the main RCT is the length (2 weeks for the pilot, 3 months for the main RCT); otherwise, they will receive the same experience. The pilot phase intends to test out a mini version of the full intervention and get participant feedback so that the study team can improve the user experience before conducting the main intervention study.

Participants in 4 of the 5 study arms will be given vouchers for use on Instacart to buy fruit and vegetables ($160 a month). They will be given an individualized link to a special study website that is an Instacart virtual store where they can order food items to be delivered. Weekly, Instacart will send us data on how much is left in terms of unexpended vouchers and what food is purchased for each study ID each month.

Initial Feasibility Test (2 Weeks): Before enrolling participants in this phase of the study, the study team will examine strategies for uptake and engagement through one rapid 10-person studies followed by semi-structured interviews to gather feedback on ways to improve the user experience. There will be a cohort of 10 participants randomized 2 in each of the 5 study arms. Each interview will be audio-recorded with permission from the participant and subsequently transcribed for analysis. Interviews will take place over the phone or on Zoom and will be recorded using an audio recorder. Audio files will be uploaded to a third-party professional transcription service, which will transcribe the recordings and send us the transcripts for analysis. Participants that sign up for their Instacart account within 48 hours will receive a $25 Instacart gift card. All participants in the intervention arms during this phase will receive $40 per week for two weeks to be used to subsidize the purchase of foods on the healthy foods list (denoted by Instacart on the virtual storefront). Participants in the control arm will receive $5 per week for two weeks to cover additional service fees, delivery fees, and driver tips. This will be done twice to reach high rates of initial enrollment and ongoing engagement. This will also test the integration of our trial platform (W2H), connection to Instacart, and receipt of data from Instacart at the individual level. These iterative studies will be used to get participant input into the user experience and to streamline our on-boarding processes. Participants will also receive $50 to debrief with the study team on their experience.

Randomized Controlled Trial (3 Months): The study team then plans to test modifying choice architecture and different ways of presenting incentives to affect the degree to which these strategies change healthy food purchasing behavior.

All participants will start in the study at the beginning of the month. If they do not complete their enrollment by the 5th day of the month, they will be paused until the 1st business day of the following month.

In the RCT phase, participants will be reached out to by text and sent to a Way to Health study link where they will be asked to first complete a brief eligibility survey via text message. Eligibility questions include whether the participant is comfortable online shopping and if they have a backup payment method for foods they purchase over and above the value of the subsidies.

Participants will complete dietary recall questionnaires at 0 and 3 months via W2H. The study team will use the Diet.ID validated a two-minute dietary assessment tool (https://www.dietid.com/). As part of the 3-month assessment, participants will be asked questions about their study experience. Participants will be compensated $25 for completing instacart sign up within 48 hours, $25 for the baseline dietary survey and $25 for completing the 3-month dietary survey and exit survey and $50 for completing a hemoglobin A1c lab after 3 months.

At the completion of the 3-month study period, a subset of participants (total of 42, selecting those with highest and lowest % of fruit and vegetable voucher use each month) will be invited to complete semi-structured exit interviews conducted by a trained research coordinator over the phone or through Zoom. Participants will receive an extra $50 for completing these interviews.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 30 and 70
* Patients in the Penn Medicine system who have obesity (BMI>or=30) and diabetes (last A1C>8 in the 90 days prior to data pull)
* Self-report being comfortable online shopping
* Have a backup payment option available to use in registering for Instacart

Exclusion Criteria:

* Not fluent in English
* Opted out of research
* The patient does not have a Primary care provider assigned
* The patient is part of a Penn primary care practice engaged with the Healthy Heart Program

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2026-03-21 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the total expenditures spent on fruits and vegetables (dollars spent inclusive of application of subsidies) | At the end of the 3 month intervention
  The primary outcome will be the total expenditures spent on fruits and vegetables (dollars spent inclusive of application of subsidies)

SECONDARY OUTCOMES:
Mean percentage of the $160 subsidy used each month in the intervention arms. | At the end of the 3 month intervention
  Secondary outcome include the mean percentage of the $160 subsidy used each month in the intervention arms.
Change in hemoglobin A1c | At the end of the 3 month intervention
  Secondary outcome include change from baseline in hemoglobin A1c.
Percentage of expenditures spent on eligible fruits and vegetables | At the end of the 3 month intervention
  percentage of expenditures spent on eligible fruits and vegetables (i.e., total spent on fruits and vegetables/total spent)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, MD,PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- The University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hua SV, Klaiman T, Coratti S, White J, John A, Putt ME, Dixon E, Posner H, Volpp KG. Using a human-centered design framework and behavioral economic interventions to increase fruit and vegetable purchases in an online grocery store: Study design and methodologies. Contemp Clin Trials. 2025 Jun;153:107921. doi: 10.1016/j.cct.2025.107921. Epub 2025 Apr 17. PMID 40252826